CLINICAL TRIAL: NCT01267253
Title: A Phase II Evaluation of Brivanib (BMS582664) in the Treatment of Persistent or Recurrent Carcinoma of the Cervix (BMS Study CA182-048)
Brief Title: Brivanib Alaninate in Treating Patients With Persistent or Recurrent Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0227G; NCI-2011-03814 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000690083; CA182-048; GOG-0227G; GOG-0227G (Other: NRG Oncology); GOG-0227G (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2010-12-24; First posted 2010-12-28 (Estimated); Results first posted 2017-01-04 (Estimated); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Cervical Adenocarcinoma; Cervical Adenosquamous Carcinoma; Cervical Squamous Cell Carcinoma, Not Otherwise Specified; Persistent Disease; Recurrent Cervical Carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — brivanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (brivanib alaninate) (Experimental): Patients receive brivanib alaninate PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Brivanib Alaninate; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Brivanib Alaninate — Given PO
  Other Names: BMS 582664; BMS-582664
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies how well brivanib alaninate works in treating patients with cervical cancer that has come back. Brivanib alaninate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth or by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the proportion of patients with persistent or recurrent cervical cancer, who survive progression-free for at least 6 months and the proportion of patients who have objective tumor response (complete or partial), treated with brivanib (brivanib alaninate).

II. To determine the nature and degree of toxicity of brivanib in this cohort of patients.

SECONDARY OBJECTIVES:

I. To estimate the progression-free survival (PFS) and overall survival (OS) of patients with persistent or recurrent cervical cancer treated with brivanib.

TERTIARY OBJECTIVES:

I. To obtain the serum expression levels of surrogate markers of brivanib effects including angiogenic factors (vascular endothelial growth factor [VEGF] and basic fibroblast growth factor [bFGF]) and markers of endothelial damage (E-selectin, vascular cell adhesion molecule 1 [VCAM-1], and (intercellular adhesion molecule 1 [ICAM-1]). (exploratory) II. To determine whether these marker expression levels alone or in combination are associated with response, PFS, or overall survival. (exploratory)

OUTLINE:

Patients receive brivanib alaninate orally (PO) once daily (QD) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have persistent or recurrent squamous cell carcinoma, adenosquamous carcinoma, adenocarcinoma, or non-squamous cell carcinoma of the cervix with documented disease progression (disease not amenable to curative therapy); histologic confirmation of the original primary tumor is required via the pathology report
* All patients must have measurable disease, defined by Response Evaluation Criteria In Solid Tumors (RECIST 1.1); measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded); each lesion must be >= 10 mm when measured by computed tomography (CT), magnetic resonance imaging (MRI) or caliper measurement by clinical exam; or >= 20 mm when measured by chest x-ray; lymph nodes must be >= 15 mm in short axis when measured by CT or MRI
* Patient must have at least one ?target lesion? to be used to assess response on this protocol as defined by RECIST 1.1

  * Tumors within a previously irradiated field will be designated as ?non-target? lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy
* Patients must not be eligible for a higher priority Gynecologic Oncology Group (GOG) protocol, if one exists

  * In general, this would refer to any active GOG phase III protocol or rare tumor protocol for the same patient population
* Patients who have received one prior regimen must have a GOG performance status of 0, 1, or 2

  * Patients who have received two prior regimens must have a GOG performance status of 0 or 1
* Recovery from effects of recent surgery, radiotherapy, or chemotherapy

  * Patients should be free of active infection requiring antibiotics (with the exception of uncomplicated urinary tract infection [UTI])
  * Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to registration
  * Any other prior therapy directed at the malignant tumor, including chemotherapy and immunologic agents, must be discontinued at least three weeks prior to registration
  * Any prior radiation therapy must be completed at least 4 weeks prior to registration
  * At least 4 weeks must have elapsed from the time of any major surgical procedure
* Patients must have had one prior systemic chemotherapeutic regimen for management of advanced, metastatic, or recurrent carcinoma of the cervix; chemotherapy administered concurrent with primary radiation (e.g.; weekly cisplatin) is not counted as a systemic chemotherapy regimen for management of advanced, metastatic, or recurrent disease; adjuvant chemotherapy given following the completion of radiation therapy (or concurrent chemotherapy and radiation therapy) is not counted as a systemic chemotherapy regimen for management of advanced, metastatic, or recurrent disease (e.g.; paclitaxel and carboplatin for up to 4 cycles)
* Patients are allowed to receive, but are not required to receive, one additional cytotoxic regimen for management of recurrent or persistent disease
* Patients must have NOT received any non-cytotoxic (biologic or targeted) agents as part of their primary treatment or for management of recurrent or persistent disease

  * Non-cytotoxic (biologic or targeted) agents include (but are not limited to) monoclonal antibodies, cytokines, and small-molecule inhibitors of signal transduction
* Absolute neutrophil count (ANC) greater than or equal to 1,500/mcl
* Platelets greater than or equal to 100,000/mcl
* Hemoglobin >= 9 g/dl
* Creatinine less than or equal to 1.5 x institutional upper limit of normal (ULN)
* Urinalysis needs to be assessed at baseline and proteinuria must be less than or equal to 2+ by dipstick

  * If the urine dipstick is > 2+, a 24-hour protein level can be done, as clinically indicated by the investigator

    * The 24-hour protein level must be less than or equal to 3.5 g/24 hours
* Bilirubin less than or equal to 1.5 x ULN
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to 3 x ULN
* Alkaline phosphatase less than or equal to 2.5 x ULN
* Albumin greater than or equal to 2.5 g/dl
* Neuropathy (sensory and motor) less than or equal to grade 1
* Prothrombin time (PT) such that international normalized ratio (INR) is =< 1.5 x ULN; patients on therapeutic warfarin are excluded from trial, anticoagulation with low molecular weight heparin is allowed
* Patients must have signed an approved informed consent and authorization permitting release of personal health information
* Patients of childbearing potential must have a negative serum pregnancy test performed 48 hours prior to study entry and be practicing an effective form of contraception during the study and for at least 3 months after receiving the final treatment of brivanib
* All patients must have a baseline electrocardiogram completed prior to study entry

  * Baseline electrocardiogram (ECG) should be repeated if corrected QT interval (QTc) is found to be > 450 msec; QTc must NOT be > 450 msec on both ECGs performed during the same visit

Exclusion Criteria:

* Patients who have had prior therapy with brivanib or anti-vascular, anti-PDGFR (platelet-derived growth factor receptor) or anti-FGFR (fibroblast growth factor receptor) therapy
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer and other specific malignancies, are excluded if there is any evidence of the other malignancy being present within the last three years; patients are also excluded if their previous cancer treatment contraindicates this protocol therapy
* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis OTHER THAN for the treatment of cervical cancer within the last three years are excluded

  * Prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease
* Patients who have received prior chemotherapy for any abdominal or pelvic tumor OTHER THAN for the treatment of cervical cancer within the last three years are excluded

  * Patients may have received prior adjuvant chemotherapy for localized breast cancer, provided that it was completed more than three years prior to registration, and that the patient remains free of recurrent or metastatic disease
* Patients that are on required chronic anti-platelet therapy (aspirin > 300 mg/day, or clopidogrel greater than or equal to 75 mg/day)
* Patients with gastrointestinal bleeding or any other hemorrhage/bleeding event >= grade 3 of the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) within 30 days prior to study entry
* Patients with a history of poor wound healing, non-healing ulcers, or bone fractures within the last 3 months
* Patients with uncontrolled or significant cardiovascular disease including any of the following:

  * Myocardial infarction within 12 months
  * Uncontrolled angina within 12 months
  * Class III-IV New York Heart Association (NYHA) congestive heart failure
  * Uncontrolled hypertension despite anti-hypertensive therapy

    * Blood pressure (BP) must be less than or equal to 140/90 at screening
    * Subjects with a history of hypertension who are receiving treatment with calcium channel blockers that are cytochrome P450 family 3, subfamily A, polypeptide 4 (CYP3A4) inhibitors should be changed to an alternative antihypertensive medication before study entry
  * History of stroke, transient ischemic attack (TIA), or other central nervous system (CNS) ischemic event
  * Cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or digoxin
  * Patients must have pre-therapy left ventricular ejection fraction (LVEF) testing and have an ejection fraction >= institutional lower limit of normal (LLN)
  * Patients with valvular heart disease >= grade 2
* Patients with a serious uncontrolled medical disorder or active infection which would impair the ability of the subject to receive protocol therapy or whose control may be jeopardized by the complications of this therapy
* Pre-existing thyroid abnormality with thyroid function that cannot be maintained in the normal range with medication
* Patients with hyponatremia (sodium < 130 mEq/L)
* Patients with active/known human immunodeficiency virus (HIV), hepatitis B, or hepatitis C; HIV-positive subjects on combination antiretroviral therapy are ineligible
* Patients with known brain metastases
* Patients who are pregnant or nursing
* Patients with inability to swallow tablets or untreated malabsorption syndrome
* Patients with baseline serum potassium < 3.5 mmol/L (potassium supplementation may be given to restore the serum potassium above this level prior to entry study)
* Patients on therapeutic warfarin anticoagulation are excluded

  * Patients converted to anticoagulation with low molecular weight heparin will be allowed provided the patient?s PT is such that INR is =< 1.5 x ULN

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-04-04 (Actual); Primary Completion 2014-02-28 (Actual); Study Completion 2014-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John K Chan, Principal Investigator — NRG Oncology
Locations (43):
- United States (43):
  - Saint Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Florida Hospital Orlando, Orlando, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Memorial Health University Medical Center, Savannah, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Sudarshan K Sharma MD Limited-Gynecologic Oncology, Hinsdale, Illinois
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Baystate Medical Center, Springfield, Massachusetts
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - CoxHealth South Hospital, Springfield, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Baylor All Saints Medical Center at Fort Worth, Fort Worth, Texas
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

REFERENCES:
- [Derived] Chan JK, Deng W, Higgins RV, Tewari KS, Bonebrake AJ, Hicks M, Gaillard S, Ramirez PT, Chafe W, Monk BJ, Aghajanian C. A phase II evaluation of brivanib in the treatment of persistent or recurrent carcinoma of the cervix: An NRG Oncology/Gynecologic Oncology Group study. Gynecol Oncol. 2017 Sep;146(3):554-559. doi: 10.1016/j.ygyno.2017.05.033. Epub 2017 Jul 18. PMID 28728751

RESULTS

PARTICIPANT FLOW:
Groups:
- Brivanib: Brivanib 800mg administered orally every day on days 1 to 28 of each cycle until disease progression or adverse effects prohibit further treatment. One cycle is 28 days.
Period: Overall Study
Arm/Group | Brivanib
Started | 31
Completed | 28 (Eligible and treated patients)
Not Completed | 3
Not completed — Ineligible - required test not done | 1
Not completed — Inevaluable-never received study treatme | 2

BASELINE CHARACTERISTICS:
Population: Eligible and treated participants
Arm/Group | Brivanib
Number analyzed (Participants) | 28
Age, Customized [Count of Participants; unit: Participants]
  30-39 years | 8
  40-49 years | 9
  50-59 years | 7
  60-69 years | 2
  70-79 years | 2
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 28
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Tumor Response
Description: Proportion of participants with objective tumor response. Objective tumor response is defined as complete or partial tumor response assessed by RECIST 1.1
Time Frame: Every other cycle for first 6 months; then every 3 months thereafter until disease progression confirmed; and at any other time if clinically indicated based on symptoms or physical signs suggestive of progressive disease.
Population: Eligible and Treated participants
Measure: Number (90% Confidence Interval); unit: proportion
Arm/Group | Brivanib
Number analyzed (Participants) | 28
proportion | 0.071 [0.02 to 1.00]

2. Primary Outcome: PFS for at Least 6 Months Without Non-protocol Therapy From Study Entry.
Description: Proportion of participants who survive progression-free for at least 6 months without non-protocol therapy from study entry. Progression is assessed by RECIST 1.1.
Time Frame: Every other cycle for first 6 months; then every 3 months therafter until disease progression confirmed; and at any other time if cliniclly indicated based on symptoms or physical signs suggestive of progressive disease
Population: Eligible and treated participants
Measure: Number (90% Confidence Interval); unit: proportion
Arm/Group | Brivanib
Number analyzed (Participants) | 28
proportion | 0.179 [0.09 to 1.00]

3. Primary Outcome: Adverse Events (Grade 3 or Higher) During Treatment Period
Description: Number of participants with a maximum grade of 3 or higher during treatment period. Adverse events are graded and categorized using CTCAE v.4.0
Time Frame: During treatment period and up to 30 days after stopping the study treatment.
Population: Eligible and Treated Participants
Measure: Number; unit: Participants
Arm/Group | Brivanib
Number analyzed (Participants) | 28
Participants
  Leukopenia | 0
  Thrombocytopenia | 0
  Neutropenia | 0
  Anemia | 4
  Other Investigations | 4
  Cardiac Disorders | 1
  Gastrointestinal Disorders | 7
  General disorders & administration site conditions | 2
  Hepatobiliary Disorders | 1
  Infections and infestations | 4
  Metabolism and nutrition disorders | 5
  Musculoskeletal & connective tissue disorders | 3
  Neoplasms benign, malignant & unspecified | 2
  Nervous system disorders | 3
  Renal and urinary disorders | 2
  Vascular Disorders | 5

4. Secondary Outcome: Progression-free Survival
Description: Progression-free survival is the period of time from study entry to time of disease progression, death or date of last contact, whichever occurs first. Progression is assessed by RECIST 1.1
Time Frame: From study entry to time of progression or death, whichever occurs first, up to 5 years of follow-up
Population: Eligible and Treated Participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Brivanib
Number analyzed (Participants) | 28
Months | 3.2 [2.0 to 4.4]

5. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the duration of time from study entry to time of death or the date of last contact..
Time Frame: From study entry to time of death or the date of last contact, up to 5 years of follow-up.
Population: Eligible and Treated Patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Brivanib
Number analyzed (Participants) | 28
Months | 7.9 [6.1 to 11.7]

6. Other Pre Specified Outcome: Serum Expression Levels of Surrogate Markers of Brivanib Alaninate Effects Including Angiogenic Factors (VEGF and bFGF) and Markers of Endothelial Damage (E-selectin, VCAM-1, and ICAM-1)
Description: Surrogate markers will be associated with response, PFS, and OS.
Time Frame: Up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) occurring during treatment and up to 30 days after stopping the study treatment are reported.
Arm/Group | Brivanib
Serious Adverse Events (participants affected / at risk) | 14/28
Other Adverse Events (participants affected / at risk) | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brivanib (N=28)
Anemia (Blood and lymphatic system disorders) | 1
Pulmonary Valve Disease (Cardiac disorders) | 1
Colonic Hemorrhage (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 1
Rectal Hemorrhage (Gastrointestinal disorders) | 1
Mucositis Oral (Gastrointestinal disorders) | 1
Bile Duct Stenosis (Hepatobiliary disorders) | 1
Sepsis (Infections and infestations) | 1
Lung Infection (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Neoplasms Benign, Malignant And Unspecified (Incl (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Reversible Posterior Leukoencephalopathy Syndrome (Nervous system disorders) | 1
Urinary Tract Obstruction (Renal and urinary disorders) | 1
Urinary Retention (Renal and urinary disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brivanib (N=28)
Anemia (Blood and lymphatic system disorders) | 23
Palpitations (Cardiac disorders) | 1
Left Ventricular Systolic Dysfunction (Cardiac disorders) | 1
Sinus Tachycardia (Cardiac disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 3
Hearing Impaired (Ear and labyrinth disorders) | 2
Hypothyroidism (Endocrine disorders) | 2
Hyperthyroidism (Endocrine disorders) | 1
Eye Disorders - Other (Eye disorders) | 1
Photophobia (Eye disorders) | 1
Blurred Vision (Eye disorders) | 2
Dysphagia (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 2
Dry Mouth (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 9
Diarrhea (Gastrointestinal disorders) | 11
Vomiting (Gastrointestinal disorders) | 15
Bloating (Gastrointestinal disorders) | 3
Abdominal Pain (Gastrointestinal disorders) | 10
Rectal Hemorrhage (Gastrointestinal disorders) | 3
Oral Dysesthesia (Gastrointestinal disorders) | 1
Mucositis Oral (Gastrointestinal disorders) | 4
Abdominal Distension (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 20
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1
Rectal Pain (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Pain (General disorders) | 5
Flu Like Symptoms (General disorders) | 1
Non-Cardiac Chest Pain (General disorders) | 3
Edema Limbs (General disorders) | 4
Fatigue (General disorders) | 22
Fever (General disorders) | 5
Chills (General disorders) | 2
Allergic Reaction (Immune system disorders) | 1
Upper Respiratory Infection (Infections and infestations) | 1
Tooth Infection (Infections and infestations) | 1
Skin Infection (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 5
Abdominal Infection (Infections and infestations) | 1
Wound Complication (Injury, poisoning and procedural complications) | 1
Bruising (Injury, poisoning and procedural complications) | 1
Weight Loss (Investigations) | 6
Weight Gain (Investigations) | 1
Platelet Count Decreased (Investigations) | 8
Lymphocyte Count Decreased (Investigations) | 5
Hemoglobin Increased (Investigations) | 1
Ejection Fraction Decreased (Investigations) | 2
Creatinine Increased (Investigations) | 4
Cardiac Troponin T Increased (Investigations) | 1
Neutrophil Count Decreased (Investigations) | 5
Blood Bilirubin Increased (Investigations) | 3
White Blood Cell Decreased (Investigations) | 12
Aspartate Aminotransferase Increased (Investigations) | 8
Alkaline Phosphatase Increased (Investigations) | 7
Alanine Aminotransferase Increased (Investigations) | 7
Hyponatremia (Metabolism and nutrition disorders) | 10
Hypomagnesemia (Metabolism and nutrition disorders) | 6
Hypokalemia (Metabolism and nutrition disorders) | 8
Hypocalcemia (Metabolism and nutrition disorders) | 8
Hypoalbuminemia (Metabolism and nutrition disorders) | 9
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 8
Hypercalcemia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 3
Anorexia (Metabolism and nutrition disorders) | 15
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 1
Joint Range Of Motion Decreased (Musculoskeletal and connective tissue disorders) | 1
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 9
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Seizure (Nervous system disorders) | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 8
Paresthesia (Nervous system disorders) | 1
Memory Impairment (Nervous system disorders) | 1
Headache (Nervous system disorders) | 11
Dizziness (Nervous system disorders) | 6
Concentration Impairment (Nervous system disorders) | 2
Aphonia (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 2
Hallucinations (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 4
Anxiety (Psychiatric disorders) | 3
Urinary Urgency (Renal and urinary disorders) | 1
Urinary Tract Obstruction (Renal and urinary disorders) | 1
Urinary Retention (Renal and urinary disorders) | 2
Urinary Incontinence (Renal and urinary disorders) | 1
Urinary Tract Pain (Renal and urinary disorders) | 4
Urinary Frequency (Renal and urinary disorders) | 6
Proteinuria (Renal and urinary disorders) | 6
Hemoglobinuria (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 3
Cystitis Noninfective (Renal and urinary disorders) | 1
Chronic Kidney Disease (Renal and urinary disorders) | 1
Reproductive System And Breast Disorders - Other (Reproductive system and breast disorders) | 1
Vaginal Pain (Reproductive system and breast disorders) | 2
Vaginal Hemorrhage (Reproductive system and breast disorders) | 1
Vaginal Dryness (Reproductive system and breast disorders) | 1
Pelvic Pain (Reproductive system and breast disorders) | 2
Vaginal Discharge (Reproductive system and breast disorders) | 2
Respiratory, Thoracic And Mediastinal Disorders - (Respiratory, thoracic and mediastinal disorders) | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 2
Skin And Subcutaneous Tissue Disorders - Other (Skin and subcutaneous tissue disorders) | 1
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Rash Acneiform (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 2
Nail Ridging (Skin and subcutaneous tissue disorders) | 1
Nail Loss (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2
Superior Vena Cava Syndrome (Vascular disorders) | 1
Lymphedema (Vascular disorders) | 2
Hypertension (Vascular disorders) | 12
Hot Flashes (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No